## J2G-MC-JZJV Statistical Analysis Plan

An Open-Label Study to Investigate the Effect of Selpercatinib on the Pharmacokinetics of Dabigatran in Healthy Volunteers

NCT04782076

Approval Date: 23-Feb-2021

## STATISTICAL ANALYSIS PLAN

# An Open-Label Study to Investigate the Effect of Selpercatinib on the Pharmacokinetics of Dabigatran in Healthy Volunteers

Statistical Analysis Plan Status: Final Statistical Analysis Plan Date: 23 February 2021

Study Drug: LY3527723

Sponsor Reference: J2G-MC-JZJV Covance CRU Study: 1000071- 8445328

Clinical Phase I

Approval Date: 23-Feb-2021 GMT

Final, 23 February 2021 

## 1. TABLE OF CONTENTS

| 1. | <b>TABLE</b> | OF CONTENTS | 2 |
|---|---|---|---|
| 2. | ABBRE | VIATIONS | 3 |
| 3. | INTROI | DUCTION | 5 |
| 4. | STUDY | OBJECTIVES AND ENDPOINTS | 5 |
| 5. | STUDY | DESIGN | 6 |
| 6. | TREAT | MENTS | 6 |
| 7. | SAMPL | E SIZE JUSTIFICATION | 7 |
| 8. | <b>DEFINI</b> | TION OF ANALYSIS POPULATIONS | 7 |
| 9. | STATIS | TICAL METHODOLOGY | 7 |
| | 9.1 Gen | eral | 7 |
| | 9.2 Den | nographics and Participant Disposition | 8 |
| | 9.3 Phan | rmacokinetic Assessment | 8 |
| | 9.3.1 | Pharmacokinetic Analysis | 8 |
| | 9.3.2 | Pharmacokinetic Statistical Methodology | . 12 |
| | 9.4 Safe | ety and Tolerability Assessments | . 12 |
| | 9.4.1 | Adverse events | . 12 |
| | 9.4.2 | Concomitant medication. | . 13 |
| | 9.4.3 | Clinical laboratory parameters | . 13 |
| | 9.4.4 | Vital signs | . 13 |
| | 9.4.5 | Electrocardiogram (ECG) | . 13 |
| | 9.4.6 | Hepatic Monitoring | . 13 |
| | 9.4.7 | Other assessments | . 15 |
| | 9.4.8 | Safety and Tolerability Statistical Methodology | . 15 |
| 10 | . INTERI | M ANALYSES | . 15 |
| 11 | . CHANG | ES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES | . 15 |
| 12 | . REFERI | ENCES | . 15 |
| 13 | . DATA F | PRESENTATION | . 15 |
| | 13.1 Derived Parameters | | |
| | 13.2 Miss | sing Data | . 16 |
| | 13.3 Insu | fficient Data for Presentation | . 16 |

#### 2. ABBREVIATIONS

Abbreviations pertain to the Statistical Analysis Plan (SAP) only (not the tables, figures and listings [TFLs]).

AE Adverse event

ALP Alkaline phosphatase

ALT Alanine aminotransferase
AST Aspartate aminotransferase

AUC Area under the concentration versus time curve

AUC $(0-\infty)$  Area under the concentration versus time curve from time zero to infinity

AUC(0- $t_{last}$ ) Area under the concentration versus time curve from time zero to time t,

where t is the last time point with a measurable concentration

BQL Below the quantifiable lower limit of the assay

CI Confidence interval

CL/F Apparent total body clearance of drug calculated after extra-vascular

administration

C<sub>max</sub> Maximum observed drug concentration

CRU Clinical Research Unit
CSR Clinical Study Report
DDI Drug-drug interaction
ECG Electrocardiogram

ICH International Conference on Harmonisation

MedDRA Medical Dictionary for Regulatory Activities

P-gp P-glycoprotein
PK Pharmacokinetic

SAE Serious adverse event
SAP Statistical Analysis Plan

SD Standard deviation

t<sub>1/2</sub> Half-life associated with the terminal rate constant ( $\lambda_z$ ) in

non-compartmental analysis

TBL Total bilirubin

TEAE Treatment-emergent adverse event

TFLs Tables, Figures, and Listings

t<sub>max</sub> Time of maximum observed drug concentration

| Statistical Analysis Plan | |
|----------------------------|-----------------|
| Covance Clinical Study No. | 1000071-8445328 |

# CONFIDENTIAL Sponsor Reference J2G-MC-JZJV

| ULN | Upper limit of normal |
|---|---|
| V <sub>ss</sub> /F | Apparent volume of distribution at steady state after extra-vascular administration |
| $V_z/F$ | Apparent volume of distribution during the terminal phase after extravascular administration |
| WHO | World Health Organization |

Final, 23 February 2021 

#### 3. INTRODUCTION

This SAP has been developed after review of the Clinical Study Protocol (final version dated 21 December 2020).

This SAP describes the planned analysis of the safety, tolerability and pharmacokinetic (PK) data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shell document.

The intent of this document is to provide guidance for the statistical and PK analyses of data. In general, the analyses are based on information from the protocol, unless they have been modified by agreement with Eli Lilly and Company. A limited amount of information concerning this study (e.g., objectives, study design) is given to help the reader's interpretation. For open-label studies, this SAP must be signed off prior to first participant visit for this study. When the SAP and TFL shells are agreed upon and finalized, they will serve as the template for this study's CSR.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified in the CSR. Any substantial deviations from this SAP will be agreed upon with Eli Lilly and Company and identified in the CSR. Any minor deviations from the TFLs may not be documented in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials<sup>1</sup> and the ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports<sup>2</sup>.

#### 4. STUDY OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the effect of selpercatinib on<br>P-glycoprotein (P-gp) activity in healthy<br>participants. | <ul> <li>Maximum observed drug concentration<br/>(C<sub>max</sub>) and area under the concentration<br/>versus time curve from time zero to<br/>infinity (AUC[0-∞]) of dabigatran to<br/>assess P-gp activity.</li> </ul> |
| Secondary | |
| To evaluate the safety and tolerability of dabigatran in combination with selpercatinib in healthy participants. | • Summary of the number of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). |
| • To evaluate the PK of selpercatinib. | • C <sub>max</sub> , AUC(0-∞), and time of maximum observed drug concentration (t <sub>max</sub> ) of selpercatinib. |

Final, 23 February 2021 

#### 5. STUDY DESIGN

This is a Phase 1, fixed-sequence, open-label study in healthy participants that will study dabigatran P-gp drug-drug interaction (DDI) with selpercatinib. The anticipated study duration for each individual participant is approximately 8 weeks.

#### Screening

All participants will be screened within 28 days prior to enrollment (Day 1).

#### Treatment and Assessment Period

Eligible participants will take part in 1 treatment period. Participants will be admitted to the clinical research unit (CRU) on Day -1 and remain resident in the CRU until discharge on Day 11. All participants will receive a single dose of 150 mg dabigatran on Day 1 and a single dose of 150 mg dabigatran coadministered with a single dose of 160 mg selpercatinib on Day 8. There will be a washout period of 7 days between dosing on Days 1 and 8.

PK blood sampling and safety assessments, including vital signs measurements, physical examinations, clinical laboratory tests, electrocardiograms (ECGs), and adverse event (AE) recording, will be performed.

#### Follow-up

Participants will return to the CRU for a safety follow-up visit within 14 to 17 days after the final dose.

The study schema is shown in Figure 1.



Figure 1: J2G-MC-JZJV Study Schema

#### 6. TREATMENTS

The following is a list of the study treatment abbreviations that will be used in the TFLs. In AE outputs, treatment labels will also contain "(Day X)" information.

Final, 23 February 2021 

| Day | Study Treatment Name | Treatment order in TFL |
|-----|------------------------------------------|------------------------|
| 1 | 150 mg dabigatran | 1 |
| 8 | 150 mg dabigatran + 160 mg selpercatinib | 2 |

#### 7. SAMPLE SIZE JUSTIFICATION



#### 8. DEFINITION OF ANALYSIS POPULATIONS

The "Entered" population will consist of all participants who signed the informed consent form.

The "Enrolled/Intent-to-Treat" population will consist of all participants assigned to treatment, regardless of whether they take any doses of study intervention, or if they take the correct treatment.

The "Safety" population will consist of all participants assigned to dabigatran, and who take at least one dose of study intervention.

The "Pharmacokinetic Analysis" population will consist of all participants who received at least one dose of dabigatran and have evaluable PK data. Participants may be excluded from the PK summary statistics and statistical analysis if a participant has an AE of vomiting that occurs at or before 2 times median t<sub>max</sub>, or 2 times individual t<sub>max</sub> if individual t<sub>max</sub> is achieved.

All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when participants are assigned to analysis populations.

#### 9. STATISTICAL METHODOLOGY

#### 9.1 General

Data listings will be provided for all data that are databased. Summary statistics and statistical analysis will only be presented for data where detailed in this SAP. For continuous data, summary statistics will include the arithmetic mean, arithmetic standard deviation (SD), median, minimum, maximum and N; for log-normal data (e.g. the PK parameters: AUCs and C<sub>max</sub>) the geometric mean and geometric coefficient of variation will also be presented. For categorical data, frequency count and percentages will be presented. Data listings will be provided for all participants up to the point of withdrawal, with any participants excluded from the relevant

population highlighted. Summary statistics and statistical analyses will generally only be performed for participants included in the relevant analysis population. For the calculation of summary statistics and statistical analysis, unrounded data will be used.

Mean change from baseline is the mean of all individual participants' change from baseline values. Each individual change from baseline will be calculated by subtracting the individual participant's baseline value from the value at the timepoint. The individual participant's change from baseline values will be used to calculate the mean change from baseline using a SAS procedure such as Proc Univariate.

Data analysis will be performed using SAS® Version 9.4 or greater.

#### 9.2 Demographics and Participant Disposition

Participant disposition will be listed. The demographic variables age, sex, race, ethnicity, country of enrolment, site ID, body weight, height and body mass index will be summarized and listed. All other demographic variables will be listed only.

#### 9.3 Pharmacokinetic Assessment

#### 9.3.1 Pharmacokinetic Analysis

Noncompartmental methods applied with a validated software program (Phoenix WinNonlin Version 8.1 or later) to the plasma concentrations of dabigatran and selpercatinib will be used to determine the following PK parameters, when possible:

| Parameter | Units | Definition |
|---|---|---|
| AUC(0-t <sub>last</sub> ) | ng.h/mL | area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration |
| $AUC(0-\infty)$ | ng.h/mL | area under the concentration versus time curve from time zero to infinity |
| $C_{max}$ | ng/mL | maximum observed drug concentration |
| $t_{max}$ | h | time of maximum observed drug concentration |
| t <sub>1/2</sub> | h | half-life associated with the terminal rate constant $(\lambda_z)$ in non-compartmental analysis |
| CL/F | L/h | apparent total body clearance of drug calculated after extra-vascular administration |
| V <sub>Z</sub> /F | L | apparent volume of distribution during the terminal phase after extra-vascular administration |
| V <sub>SS</sub> /F | L | apparent volume of distribution at steady state after extra-vascular administration |

Additional PK parameters may be calculated, as appropriate.

The software and version used for the final analyses will be specified in the CSR. Any exceptions or special handling of data will be clearly documented within the CSR.

Formatting of tables, figures and abbreviations will follow the Eli Lilly Global PK/PD/TS Tool: NON-COMPARTMENTAL PHARMACOKINETIC STYLE GUIDE. The version of the tool effective at the time of PK analysis will be followed.

#### **General PK Parameter Rules**

- Actual sampling times will be used in the final analyses of individual PK parameters, except for non-bolus pre-dose sampling times which will be set to zero.
- The  $C_{max}$  and  $t_{max}$  will be reported from observed values. If  $C_{max}$  occurs at more than one timepoint,  $t_{max}$  will be assigned to the first occurrence of  $C_{max}$ .
- The AUC parameters will be calculated using a combination of the linear and logarithmic trapezoidal methods (linear-log trapezoidal rule). The linear trapezoidal method will be applied up to t<sub>max</sub> and then the logarithmic trapezoidal method will be used after t<sub>max</sub>. The minimum requirement for the calculation of AUC will be the inclusion of at least three consecutive plasma concentrations above the lower limit of quantification, with at least one of these concentrations following C<sub>max</sub>.
- The t<sub>1/2</sub> will be calculated, when appropriate, based on the apparent terminal log-linear portion of the concentration-time curve. The start of the terminal elimination phase for each participant will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in plasma concentrations. Half-life will only be calculated when a reliable estimate for this parameter can be obtained comprising of at least 3 data points. If t<sub>1/2</sub> is estimated over a time window of less than 2 half-lives, the values will be flagged in the data listings. Any t<sub>1/2</sub> value excluded from summary statistics will be documented in the footnote of the summary table.
- A uniform weighting scheme will be used in the regression analysis of the terminal loglinear portion of the concentration-time curve.
- The parameters based on predicted last quantifiable drug concentration will be reported.

#### **Individual PK Parameter Rules**

- Only quantifiable concentrations will be used to calculate PK parameters with the exception of special handling of certain concentrations reported below the lower limit of quantitation (BQL). Plasma concentrations reported as BQL will be set to a value of zero when all of the following conditions are met:
  - The compound is non-endogenous.
  - The samples are from the initial dose period for a participant or from a subsequent dose period following a suitable wash-out period.
  - The time points occur before the first quantifiable concentration.

- All other BQL concentrations that do not meet the above criteria will be set to missing.
- Also, where two or more consecutive concentrations are BQL towards the end of a profile, the profile will be deemed to have terminated and therefore any further quantifiable concentrations will be set to missing for the calculation of the PK parameters unless it is considered to be a true characteristic of the profile of the drug.

#### **Individual Concentration vs. Time Profiles**

- Individual concentrations will be plotted utilizing actual sampling times.
- The terminal point selections will be indicated on a semi-logarithmic plot.

#### **Average Concentration vs. Time Profiles**

- The average concentration profiles will be graphed using scheduled (nominal) sampling times.
- The average concentration profiles will be graphed using arithmetic average concentrations.
- The pre-dose average concentration for single-dose data from non-endogenous compounds will be set to zero. Otherwise, only quantifiable concentrations will be used to calculate average concentrations.
- Concentrations at a sampling time exceeding the sampling time window specified in the protocol, or ± 10%, will be excluded from the average concentration profiles.
- Concentrations excluded from the mean calculation will be documented in the CSR.
- A concentration average will be plotted for a given sampling time only if 2/3 of the individual data at the time point have quantifiable measurements that are within the sampling time window specified in the protocol or ± 10%. An average concentration estimated with less than 2/3 but more than 3 data points may be displayed on the mean concentration plot if determined to be appropriate and will be documented within the CSR.

#### **Treatment of Outliers during Pharmacokinetic Analysis**

Application of this procedure to all PK analyses is not a requirement. Rather, this procedure provides justification for exclusion of data when scientifically appropriate. This procedure describes the methodology for identifying an individual value as an outlier for potential exclusion, but does not require that the value be excluded from analysis. The following methodology will not be used to exclude complete profiles from analysis.

#### Data within an Individual Profile

A value within an individual profile may be excluded from analysis if any of the following criteria are met:

- For PK profiles during multiple dosing, the concentration of the pre-dose sample exceeds all measured concentrations for that individual in the subsequent post-dose samples.
- For PK profiles during single dosing of non-endogenous compounds, the concentration in a pre-dose sample is quantifiable.
- For any questionable datum that does not satisfy the above criteria, the profile will be evaluated and results reported with and without the suspected datum.

#### Data between Individual Profiles

- 1. If n<6, then the dataset is too small to conduct a reliable range test. Data will be analyzed with and without the atypical value, and both sets of results will be reported.
- 2. If n≥6, then an objective outlier test will be used to compare the atypical value to other values included in that calculation:
  - a. Transform all values in the calculation to the logarithmic domain.
  - b. Find the most extreme value from the arithmetic mean of the log transformed values and exclude that value from the dataset.
  - c. Calculate the lower and upper bounds of the range defined by the arithmetic mean  $\pm 3*SD$  of the remaining log-transformed values.
  - d. If the extreme value is within the range of arithmetic mean  $\pm 3*SD$ , then it is not an outlier and will be retained in the dataset.
  - e. If the extreme value is outside the range of arithmetic mean  $\pm 3*SD$ , then it is an outlier and will be excluded from analysis.

If the remaining dataset contains another atypical datum suspected to be an outlier and  $n \ge 6$  following the exclusion, then repeat step 2 above. This evaluation may be repeated as many times as necessary, excluding only one suspected outlier in each iteration, until all data remaining in the dataset fall within the range of arithmetic mean  $\pm 3*SD$  of the log-transformed values.

#### Reporting of Excluded Values

Individual values excluded as outliers will be documented in the CSR. Approval of the CSR will connote approval of the exclusion.

Final, 23 February 2021 

#### 9.3.2 Pharmacokinetic Statistical Methodology



PK parameters will be summarized using descriptive statistics.

#### 9.4 Safety and Tolerability Assessments

#### 9.4.1 Adverse events

Where changes in severity are recorded in the case report form, each separate severity of the AE will be reported in the listings, only the most severe will be used in the summary tables. A pre-existing condition is defined as an AE that starts before the participant has provided written informed consent and is ongoing at consent. A non-treatment emergent AE is defined as an AE which starts after informed consent but prior to dosing. A TEAE is defined as an AE which occurs postdose or which is present prior to dosing and becomes more severe postdose.

All AEs will be listed. All TEAEs will be summarized by treatment, severity and relationship to the investigational product. The frequency (the number of AEs, the number of participants experiencing an AE and the percentage of participants experiencing an AE) of TEAEs will be

Final, 23 February 2021 

summarized by treatment, Medical Dictionary for Regulatory Activities (MedDRA) version 23.1 system organ class and preferred term. The summary and frequency AE tables will be presented for all causalities and those considered related to the investigational product by the investigator. Any SAEs will be listed, including investigational-product related SAEs.

Discontinuations due to AEs will be listed.

#### 9.4.2 Concomitant medication

Concomitant medication will be coded using the World Health Organization (WHO) drug dictionary (Version WHODDSEP20B3), and listed.

#### 9.4.3 Clinical laboratory parameters

Liver enzyme tests data (ALP, AST, ALT) will be summarized. All clinical chemistry, hematology, and urinalysis data will be listed. Additionally, clinical chemistry, hematology and urinalysis data outside the reference ranges will be listed and flagged on individual participant data listings.

#### 9.4.4 Vital signs

Vital signs data will be summarized by treatment together with changes from baseline. Baseline is defined as Day 1 predose for the first dose, and Day 7 predose for the second dose. Figures of mean vital signs and mean changes from baseline profiles will be presented by treatment, for the first 24 hours after dosing in each treatment period.

Values for individual participants will be listed.

#### 9.4.5 Electrocardiogram (ECG)

ECGs will be performed for safety monitoring purposes only and will not be presented. Any clinically significant findings from ECGs will be reported as an AE.

#### 9.4.6 Hepatic Monitoring

#### Close hepatic monitoring

If a participant who had normal or near normal baseline alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin (TBL) (i.e., <1.5× upper limit of normal [ULN]), experiences elevated ALT≥3× ULN, AST≥3× ULN, ALP≥2× ULN, or TBL≥2× ULN, laboratory tests should be repeated within 48 to 72 hours, including ALT, AST, ALP, TBL, direct bilirubin, gamma-glutamyltransferase, and creatinine kinase to confirm the abnormality and to determine if it is increasing or decreasing.

In participants enrolled with elevated baseline ALT, AST, ALP or TBL ( $\geq 1.5 \times$  ULN), the thresholds for close monitoring are ALT $\geq 2 \times$  baseline, AST $\geq 2 \times$  baseline, ALP $\geq 2 \times$  baseline, or TBL $\geq 2 \times$  baseline.

Final, 23 February 2021 

At a minimum, this evaluation should include physical examination and a thorough medical history, including symptoms, recent illnesses, (for example, heart failure, systemic infection, hypotension, or seizures), recent travel, history of concomitant medications (including over-the-counter), herbal and dietary supplements, history of alcohol drinking and other substance abuse.

If the abnormality persists or worsens, clinical and laboratory monitoring, and evaluation for possible causes of abnormal liver tests should be initiated by the investigator in consultation with the Lilly-designated medical monitor.

#### Comprehensive hepatic evaluation

If a study participant, who had baseline ALT, AST, ALP, TBL<1.5× ULN, experiences elevated ALT $\geq$ 5× ULN, AST $\geq$ 5× ULN, ALP $\geq$ 3× ULN, TBL $\geq$ 2× ULN, or elevated ALT, AST $\geq$ 3× ULN with hepatic signs/symptoms (severe fatigue, nausea, vomiting, right upper quadrant abdominal pain, fever, rash, and/or eosinophilia>5%), a comprehensive evaluation should be performed to search for possible causes of liver injury.

In participants who had elevated baseline ALT, AST, ALP, or TBL ( $\geq 1.5 \times$  ULN), the thresholds for performing this evaluation are ALT $\geq 3 \times$  baseline, AST $\geq 3 \times$  baseline, ALP $\geq 2 \times$  baseline, TBL $\geq 1.5 \times$  baseline, or ALT, AST  $\geq 2 \times$  baseline with hepatic signs/symptoms.

At a minimum, this evaluation should include physical examination and a thorough medical history, as outlined above, as well as tests for prothrombin time-international normalized ratio, viral hepatitis A, B, C, E, tests for autoimmune hepatitis, and an abdominal imaging study (for example, ultrasound or computed tomography scan).

## Additional hepatic data collection in participants who have abnormal liver tests during the study

Additional hepatic safety data collection should be performed in participants who meet 1 or more of the following 5 conditions:

- 1. Elevation of serum ALT to  $\geq$ 5× ULN on 2 or more consecutive blood tests (if baseline ALT<1.5x ULN)
  - ➤ In participants with baseline ALT≥1.5× ULN, the threshold is ALT≥3x baseline on 2 or more consecutive tests
- 2. Elevation of TBL to  $\geq 2 \times$  ULN (if baseline TBL  $\leq 1.5 \times$  ULN)
  - ➤ In participants with baseline TBL  $\ge 1.5 \times$  ULN, the threshold should be TBL  $\ge 2x$  baseline
- 3. Elevation of serum ALP to  $\ge 2 \times$  ULN on 2 or more consecutive blood tests (if baseline ALP <1.5× ULN)
  - ➤ In participants with baseline ALP≥1.5× ULN, the threshold is ALP ≥2× baseline on 2 or more consecutive blood tests
- 4. Hepatic event considered to be an SAE

Final, 23 February 2021 

5. Discontinuation of the investigational product due to a hepatic event.

Where applicable, the following will be presented. The participants' liver disease history and associated person liver disease history data will be listed. Any concomitant medications that have potential for hepatotoxicity, including acetaminophen will be listed. Results from any hepatic monitoring procedures, such as a magnetic resonance elastography scan, and biopsy assessments will be listed, if performed.

Hepatic risk factor assessment data will be listed. Liver related signs and symptoms data will be summarized by treatment and listed. Alcohol and recreational drug use data will also be listed.

All hepatic chemistry, hematology, coagulation, and serology data will be listed. Values outside the reference ranges will be flagged on the individual participant data listings.

#### 9.4.7 Other assessments

All other safety assessments not detailed in this section will be listed but not summarized or statistically analyzed.

#### 9.4.8 Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

#### 10. INTERIM ANALYSES

No interim statistical analyses are planned.

#### 11. CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES

There were no changes from the protocol specified statistical analyses.

#### 12. REFERENCES

- 1. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Statistical Principles for Clinical Trials (E9), 5 February 1998.
- 2. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Structure and Content of Clinical Study Reports (E3), 30 November 1995.

#### 13. DATA PRESENTATION

#### 13.1 Derived Parameters

Individual derived parameters (e.g. PK parameters) and appropriate summary statistics will be reported to three significant figures. Observed concentration data, e.g. C<sub>max</sub>, should be reported as received. Observed time data, e.g. t<sub>max</sub>, should be reported as received. N and percentage

Final, 23 February 2021 

values should be reported as whole numbers. Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

### 13.2 Missing Data

Missing data will not be displayed in listings.

#### 13.3 Insufficient Data for Presentation

Some of the TFLs may not have sufficient numbers of participants or data for presentation. If this occurs, the blank TFL shell will be presented with a message printed in the center of the table, such as, "No serious adverse events occurred for this study."

Final, 23 February 2021 

#### Leo Document ID = b42690b5-c820-4d21-90cb-756326f84aa4

Approver: PPD

Approval Date & Time: 23-Feb-2021 13:46:04 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 23-Feb-2021 13:49:02 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 23-Feb-2021 15:21:35 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 23-Feb-2021 15:30:36 GMT

Signature meaning: Approved